CLINICAL TRIAL: NCT00233701
Title: Normal Pressure Hydrocephalus (NPH) Registry
Status: Completed | Type: Observational
Sponsor: Codman & Shurtleff (Industry)
Collaborators: American Association of Neurological Surgeons (Other)
Responsible Party: Michael Ward, Worldwide Director, Clinical Research, Codman & Shurtleff
Other Study IDs: NPH-US04-001
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2008-10

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: NPH; Hydrocephalus
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Hydrocephalus

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall aim of the registry is to develop a longitudinal, observational database that is focused on adult patients with Normal Pressure Hydrocephalus (NPH) that can be used as a source of clinical information for individual surgeons, as well as a national data repository for scientific inquiry and publications.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational database to collect data on the characteristics, management practices, and patient outcomes of NPH patients. It will be offered to a geographically representative group of U.S. physicians who will enroll NPH patients. The physician makes his/her own clinical decisions; thus, the data captured provides current practice patterns related to diagnosis, management, and results. The registry may also assist physicians in patient follow-up and certain practice management tasks. The data collected will serve to inform the medical community on optimal care for this patient population

ELIGIBILITY:
Inclusion Criteria:

* Patient meets the diagnosis criteria for Normal Pressure Hydrocephalus
* Patient is a candidate for a hydrocephalus shunt system, per the discretion of the investigator
* Patient or legal representative has signed an informed consent form. Competency to sign the consent form will be left up to the discretion of the investigator

Exclusion Criteria:

* Patient is under the age of 18 years
* Patient has a known contraindication for a shunt
* Patient has an expected life span of less than 24 months
* Patient has an unwillingness or inability to return for required follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NPH patient who is a candidate for a shunt. Can not be under that age of 18, have a known contraindication for a shunt, or have an expected life span of less than 24 months.
Sampling Method: Non-Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2004-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Database to describe the population of patients with NPH presenting for treatment (assessed at baseline/no safety assessment) | End of trial

SECONDARY OUTCOMES:
To determine frequency of the various treatments for NPH and the outcomes of those treatment (assessed during surgery and at follow-up/no safety assessment) | End of trial

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Marmarou, Ph.D., Study Chair — Virginia Commonwealth University
Locations (28):
- United States (28):
  - Phoenix, Arizona
  - Los Angeles, California
  - Boulder, Colorado
  - Jacksonville, Florida
  - Macon, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Iowa City, Iowa
  - Lexington, Kentucky
  - Detroit, Michigan
  - Camden, New Jersey
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Youngstown, Ohio
  - Midwest City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Abington, Pennsylvania
  - Hershey, Pennsylvania
  - Johnson, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Kingsport, Tennessee
  - Dallas, Texas
  - Wichita Falls, Texas
  - Payson, Utah
  - Salt Lake City, Utah
  - Richmond, Virginia
  - La Crosse, Wisconsin

REFERENCES:
- See also: Related Info — http://www.lifenph.com